CLINICAL TRIAL: NCT01337947
Title: The Impact of Fitness on Vascular Dysfunction in Adolescents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Eugene Barrett, Eugene Barrett, MD, PhD, University of Virginia
Other Study IDs: IRB- HSR #15312
Record Dates: First submitted 2011-04-14; First posted 2011-04-19 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2011-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; adolescents; exercise; vascular function
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — perflutren

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- exercise training: 12 weeks of exercise treatment/program for DM1 subjects
  Interventions: Drug: Definity microbubbles

INTERVENTIONS:
Drug: Definity microbubbles — Definity microbubbles are used as a contrast agent to image blood flow in skeletal muscle
  Other Names: Definity

SUMMARY:
The principal hypothesis of this study is that the micro and macro vasculature of young diabetes mellitus type 1 (DM1) patients is particularly susceptible to atherogenic factors which cause vascular dysfunction at multiple levels of the arterial vasculature and that this dysfunction is demonstrable using state-of-the-art ultrasound methods. The investigators further hypothesize that interventions, such as exercise, that are readily integrated into the daily life of individuals with DM1 can mitigate or reverse these early vascular changes and thereby diminish the otherwise predictable longer-term development of cardiovascular disease (CVD) in type 1 DM

ELIGIBILITY:
Inclusion Criteria: You may be eligible if you are:

* Male or female, 12-18 years of age
* Healthy, no chronic illness other than DM1
* No medications that would affect the blood vessels
* Non-smoker
* Normal height and weight

Requirements for both groups (study 1)

* Two outpatient visits lasting ~1 to 1 ½ hours
* 1 outpatient admission lasting ~ 10 hrs
* Most visits require blood draws Requirements for second part of study for DM1 group (study 2)
* Two additional outpatient visits (one requires blood draw)
* 12 weeks of an exercise program (5 days per week, 3 of them here at UVA)
* Maintain healthy diet for those 12 weeks-you will have diet instruction
* Repeat outpatient admission as described above

Exclusion Criteria:

* under 12 or over 18 years of age
* medication that could affect the blood vessels
* smoker
* above average BMI
* chronic illness other than DM1

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: DM1 and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
arterial vascular stiffness | 2 years
  Arterial Stiffness will be measured as follows:
  1. Pulse wave velocity (m/sec)
  2. Augmentation index ( %)

SECONDARY OUTCOMES:
nitric oxide dependent vasodilation | 2 years
  NO dependent vasodilation will be measured by:
  1. Flow Mediated dilation of brachial artery (% of brachial artery diameter change)
  2. Post ischemic flow velocity in brachial artery ( m/sec)
  3. Forearm microvascular perfusion using contrast ultrasound ( video intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Barrett, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Libby P, Nathan DM, Abraham K, Brunzell JD, Fradkin JE, Haffner SM, Hsueh W, Rewers M, Roberts BT, Savage PJ, Skarlatos S, Wassef M, Rabadan-Diehl C; National Heart, Lung, and Blood Institute; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Report of the National Heart, Lung, and Blood Institute-National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Circulation. 2005 Jun 28;111(25):3489-93. doi: 10.1161/CIRCULATIONAHA.104.529651. No abstract available. PMID 15983263
- [Background] Soedamah-Muthu SS, Fuller JH, Mulnier HE, Raleigh VS, Lawrenson RA, Colhoun HM. High risk of cardiovascular disease in patients with type 1 diabetes in the U.K.: a cohort study using the general practice research database. Diabetes Care. 2006 Apr;29(4):798-804. doi: 10.2337/diacare.29.04.06.dc05-1433. PMID 16567818
- [Background] Brown A, Reynolds LR, Bruemmer D. Intensive glycemic control and cardiovascular disease: an update. Nat Rev Cardiol. 2010 Jul;7(7):369-75. doi: 10.1038/nrcardio.2010.35. Epub 2010 Apr 20. PMID 20404853
- [Background] Mahmud FH, Van Uum S, Kanji N, Thiessen-Philbrook H, Clarson CL. Impaired endothelial function in adolescents with type 1 diabetes mellitus. J Pediatr. 2008 Apr;152(4):557-62. doi: 10.1016/j.jpeds.2007.08.044. Epub 2007 Nov 5. PMID 18346515
- [Background] Devaraj S, Cheung AT, Jialal I, Griffen SC, Nguyen D, Glaser N, Aoki T. Evidence of increased inflammation and microcirculatory abnormalities in patients with type 1 diabetes and their role in microvascular complications. Diabetes. 2007 Nov;56(11):2790-6. doi: 10.2337/db07-0784. Epub 2007 Aug 8. PMID 17686944
- [Background] Jarvisalo MJ, Jartti L, Nanto-Salonen K, Irjala K, Ronnemaa T, Hartiala JJ, Celermajer DS, Raitakari OT. Increased aortic intima-media thickness: a marker of preclinical atherosclerosis in high-risk children. Circulation. 2001 Dec 11;104(24):2943-7. doi: 10.1161/hc4901.100522. PMID 11739310
- [Background] Galkina E, Ley K. Immune and inflammatory mechanisms of atherosclerosis (*). Annu Rev Immunol. 2009;27:165-97. doi: 10.1146/annurev.immunol.021908.132620. PMID 19302038
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Heitzer T, Schlinzig T, Krohn K, Meinertz T, Munzel T. Endothelial dysfunction, oxidative stress, and risk of cardiovascular events in patients with coronary artery disease. Circulation. 2001 Nov 27;104(22):2673-8. doi: 10.1161/hc4601.099485. PMID 11723017
- [Background] Fichtlscherer S, Breuer S, Zeiher AM. Prognostic value of systemic endothelial dysfunction in patients with acute coronary syndromes: further evidence for the existence of the "vulnerable" patient. Circulation. 2004 Oct 5;110(14):1926-32. doi: 10.1161/01.CIR.0000143378.58099.8C. Epub 2004 Sep 27. PMID 15451794
- [Background] Vincent MA, Clerk LH, Lindner JR, Price WJ, Jahn LA, Leong-Poi H, Barrett EJ. Mixed meal and light exercise each recruit muscle capillaries in healthy humans. Am J Physiol Endocrinol Metab. 2006 Jun;290(6):E1191-7. doi: 10.1152/ajpendo.00497.2005. PMID 16682488
- [Background] Keske MA, Clerk LH, Price WJ, Jahn LA, Barrett EJ. Obesity blunts microvascular recruitment in human forearm muscle after a mixed meal. Diabetes Care. 2009 Sep;32(9):1672-7. doi: 10.2337/dc09-0206. Epub 2009 Jun 1. PMID 19487636
- [Background] Nadeau KJ, Regensteiner JG, Bauer TA, Brown MS, Dorosz JL, Hull A, Zeitler P, Draznin B, Reusch JE. Insulin resistance in adolescents with type 1 diabetes and its relationship to cardiovascular function. J Clin Endocrinol Metab. 2010 Feb;95(2):513-21. doi: 10.1210/jc.2009-1756. Epub 2009 Nov 13. PMID 19915016
- [Background] Woo KS, Chook P, Yu CW, Sung RY, Qiao M, Leung SS, Lam CW, Metreweli C, Celermajer DS. Effects of diet and exercise on obesity-related vascular dysfunction in children. Circulation. 2004 Apr 27;109(16):1981-6. doi: 10.1161/01.CIR.0000126599.47470.BE. Epub 2004 Apr 5. PMID 15066949
- [Background] Selvin E, Bolen S, Yeh HC, Wiley C, Wilson LM, Marinopoulos SS, Feldman L, Vassy J, Wilson R, Bass EB, Brancati FL. Cardiovascular outcomes in trials of oral diabetes medications: a systematic review. Arch Intern Med. 2008 Oct 27;168(19):2070-80. doi: 10.1001/archinte.168.19.2070. PMID 18955635
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- See also: Related Info — http://www.jdrf.org